CLINICAL TRIAL: NCT01551732
Title: Anger Control Therapy (ACT) With RAGE-Control: An Outpatient Videogame-assisted Therapy for the Treatment of Anger
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gonzalez-Heydrich, Joseph, M.D. (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P00000440
Record Dates: First submitted 2011-08-31; First posted 2012-03-13 (Estimated); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Anger; Aggression
Keywords: Anger; Aggression; Biofeedback; Videogame
MeSH Terms: conditions — Aggression | interventions — Biofeedback, Psychology

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anger Control Therapy (Active Comparator): 10 session manualized cognitive behavioral anger control therapy
  Interventions: Behavioral: ACT
- ACT with RAGE-Control (Experimental): 10 session manualized cognitive behavioral anger control therapy augmented with an interactive biofeedback videogame.
  Interventions: Behavioral: ACT with RAGE-Control

INTERVENTIONS:
Behavioral: ACT — 10 session manualized cognitive behavioral anger control therapy
  Other Names: CBT
  Arms: Anger Control Therapy
Behavioral: ACT with RAGE-Control — 10 session manualized cognitive behavioral anger control therapy augmented with interactive biofeedback videogame.
  Other Names: CBT and biofeedback
  Arms: ACT with RAGE-Control

SUMMARY:
The purpose of this study is to determine whether adding an interactive biofeedback video game to anger control cognitive behavioral therapy is an effective and feasible treatment.

DETAILED DESCRIPTION:
Current treatments for pathological anger and aggression in youth are lacking in their effectiveness to motivate and engage patients in treatment. As a result, mental health providers encounter challenges due to the limited generalizability of treatment effects to real-world situations outside of the therapist's office. When behavioral treatments fail to show lasting results, children and adolescents are often placed on antipsychotic medication to control their behaviors, which may result in significant toxicity levels and for which there is limited knowledge of the long-term effects on pediatric growth and development. This study tests an interactive biofeedback video game called RAGE-Control (for Regulate and Gain Emotional-Control) as a treatment for youth exhibiting anger and aggression. Treatment with RAGE-Control seeks to motivate children and adolescents to learn and practice coping skills taught in therapy within the environment of a fun and enjoyable video game. The game provides patients a venue to practice self-regulation techniques in response to the increasing stress of the game. Providing patients with the opportunity to refine their self-regulation skills in a fast-paced challenging game is hypothesized to result in greater generalization of therapeutic skills to situations outside of the therapist's office. The goal of the treatment is to decrease patients' feelings of anger, and to increase the patients' levels of control in their emotional and behavioral responses.

ELIGIBILITY:
Inclusion Criteria:

* Ages 10 to17 years old (inclusive).
* STAXI-CA score >15 on the Trait Anger subscales.

Exclusion Criteria:

* Inability to consent, comprehend, or effectively participate in the study.
* Cognitive impairment, defined as IQ < 75.
* Change in mood stabilizing and/or anti-psychotic medication dose within 4 weeks of beginning the study or anticipation of medication changes during the study period (10 weeks).

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2011-08-31 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
State Trait Anger Expression Inventory - Child and Adolescent | Baseline and two weeks Post treatment
  This is a 35 item self-report measure of patients' subjective feelings of anger and aggression administered at the baseline assessment prior to the first session and again two weeks post treatment.

SECONDARY OUTCOMES:
Disruptive Behavior Disorder Rating Scale (DBDRS) | Baseline and two weeks post treatment
  This is an interview conducted by an investigator who is blinded to the patient's treatment assignment. The investigator conducts this interview with the patient's parent/ guardian at baseline prior to the first session and again two weeks post treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph W Gonzalez-Heydrich, MD, Study Director — Boston Children's Hospital
Locations (1):
- Joseph Gonzalez-Heydrich, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Ducharme P, Kahn J, Vaudreuil C, Gusman M, Waber D, Ross A, Rotenberg A, Rober A, Kimball K, Peechatka AL, Gonzalez-Heydrich J. A "Proof of Concept" Randomized Controlled Trial of a Video Game Requiring Emotional Regulation to Augment Anger Control Training. Front Psychiatry. 2021 Sep 1;12:591906. doi: 10.3389/fpsyt.2021.591906. eCollection 2021. PMID 34539455